CLINICAL TRIAL: NCT00374491
Title: The Long-term Degradation Outcome of Bilok Biodegradable Interference Fixation Screws Used for Bone-Patellar Tendon-Bone ACL Reconstruction
Brief Title: The Long-term Degradation Outcome of Bilok Screws Used for ACL Reconstruction
Status: Withdrawn | Type: Observational
Sponsor: ArthroCare Corporation (Other)
Other Study IDs: A0506JM; 20061028
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Anterior Cruciate Ligament
Keywords: ACL; Bone Screw; Knee

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to evaluate the long term outcome of a poly L-lactic acid / β-tricalcium phosphate (BILOK) biodegradable interference fixation screw used for arthroscopic bone-patellar tendon-bone ACL reconstruction,to determine if these BILOK screws completely biodegrade as expected three years after implantation, and to determine whether there is bone ingrowth into the defect remaining after resorption of the BILOK screw.

DETAILED DESCRIPTION:
BILOK screws have been used for ACL interference fixation in the US since the late 1990s. As yet, there are no long-term studies to demonstrate the eventual biologic outcome of these devices. Animal studies indicate that the material used in BILOK implants completely degrades after 3 years, but these reports do not indicate what takes their place. Reports of other screw materials indicate that pure PLLA screws remain intact and can be removed whole at revision surgery in the first few months to years after implantation. Recently a report of a biopsy at 2 years after surgery indicated that whole fragments of a PLLA screw were observed. Schwach and Vert suggested that a PDLLA screw (combination of dextro and levo stereoisomers) completely degrade and is replaced by bone 3 years after surgery in sheep but no information is available for the human. In addition to being limited and anecdotal, most studies evaluating the degradation of biodegradable screws used in humans are conducted using plain radiographs and MRI to evaluate the status of the biodegradable screws. A report by Bach et al evaluated the MRI appearance of a biodegradable interference screw composed of a different polymer (polyglycolic acid 67% and trimethylene carbonate 33%) in eight patients at 2 years. It showed the reabsorption of the screw but suggested that MRI is not the most effective method for determining the bone ingrowth status in the area of the resorbed screws. CT scanning is a better methodology than MRI for this application and was recently used to study the disappearance of a pure PLLA screw at least 7 years after implantation. The purpose of this study is to evaluate the long-term resorption status of a Bilok screw and determine, using CT scan, what material replaces the screw.

ELIGIBILITY:
Inclusion Criteria:

* Prior patellar tendon autograft ACL reconstruction that used poly L-lactic acid (BILOK) interference fixation screws.
* Minimum follow-up of 3 years after the index surgery.
* Subject must be able to understand the verbiage of the consent form.
* The subject must be willing to undergo a physical examination of the previously operated knee.
* The subject must be willing to undergo a radiographic examination of the previously operated knee.
* The subject must be willing to undergo a CT scan examination of the previously operated knee.
* The subject signs the IRB-approved informed consent form.
* The subject is willing and able to complete required follow-up.

Exclusion Criteria:

* Subsequent ACL surgery or bone procedures in the area of the ACL graft attachments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: F. Alan Barber, MD, Principal Investigator

REFERENCES:
- [Background] Barber FA, Elrod BF, McGuire DA, Paulos LE. Preliminary results of an absorbable interference screw. Arthroscopy. 1995 Oct;11(5):537-48. doi: 10.1016/0749-8063(95)90129-9. PMID 8534294
- [Background] Athanasiou KA, Agrawal CM, Barber FA, Burkhart SS. Orthopaedic applications for PLA-PGA biodegradable polymers. Arthroscopy. 1998 Oct;14(7):726-37. doi: 10.1016/s0749-8063(98)70099-4. PMID 9788368
- [Background] McGuire DA, Barber FA, Elrod BF, Paulos LE. Bioabsorbable interference screws for graft fixation in anterior cruciate ligament reconstruction. Arthroscopy. 1999 Jul-Aug;15(5):463-73. doi: 10.1053/ar.1999.v15.015046001. PMID 10424549
- [Background] Barber FA, Elrod BF, McGuire DA, Paulos LE. Bioscrew fixation of patellar tendon autografts. Biomaterials. 2000 Dec;21(24):2623-9. doi: 10.1016/s0142-9612(00)00130-7. PMID 11071612
- [Background] Fankhauser F, Passler JM, Schippinger G, Boldin C, Scarpatetti M. Tendon-to-bone healing of a quadrupled hamstring tendon graft fixed with biodegradable screws in an immature athlete: a radiologic, arthroscopic, histologic, and electromicroscopic investigation. Arthroscopy. 2004 Nov;20(9):992-7. doi: 10.1016/j.arthro.2004.08.007. PMID 15525934
- [Background] Schwach G, Vert M. In vitro and in vivo degradation of lactic acid-based interference screws used in cruciate ligament reconstruction. Int J Biol Macromol. 1999 Jun-Jul;25(1-3):283-91. doi: 10.1016/s0141-8130(99)00043-4. PMID 10416676
- [Background] Bach FD, Carlier RY, Elis JB, Mompoint DM, Feydy A, Judet O, Beaufils P, Vallee C. Anterior cruciate ligament reconstruction with bioabsorbable polyglycolic acid interference screws: MR imaging follow-up. Radiology. 2002 Nov;225(2):541-50. doi: 10.1148/radiol.2252010357. PMID 12409593
- [Background] Fink C, Benedetto KP, Hackl W, Hoser C, Freund MC, Rieger M. Bioabsorbable polyglyconate interference screw fixation in anterior cruciate ligament reconstruction: a prospective computed tomography-controlled study. Arthroscopy. 2000 Jul-Aug;16(5):491-8. doi: 10.1053/jars.2000.4633. PMID 10882444